CLINICAL TRIAL: NCT02165280
Title: Guided IMagery and Patient Satisfaction Following Urogynecological Surgery
Brief Title: Guided IMagery and Patient Satisfaction (GIMPS) Following Urogynecological Surgery
Acronym: GIMPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Elizabeth Mueller, M.D. Assistant Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 206481
Record Dates: First submitted 2014-06-05; First posted 2014-06-17 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic Organ Prolapse; Surgery
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Guided IMagery (GIM) (Active Comparator): If randomized to GIM, they will then be given an audio Compact Disc. Patients will be instructed to listen to the recording least once per day in a calm location during the week leading up to surgery. They will then be seen prior to surgery in the surgical waiting area where they will evaluated for anxiety, preparedness and study compliance.
  Interventions: Behavioral: Guided IMagery (GIM)
- Standard of Care (SOC) (No Intervention): Each participant will complete a baseline set of questionnaires. The Pelvic Floor Distress Inventory (PFDI) is a 20 question self-administered questionnaire on the presence and both of pelvic floor symptoms .
  The Pelvic Organ Prolapse Quantification System (POPQ) measures the topography of the vagina and is considered to be gold standard for quantifying prolapse .
  The State-Trait Anxiety Inventory (STAI) has been used extensively in research and clinical practice since its introduction in 1966 and is the most widely cited measure of anxiety.
  New measurements at the 6-week follow-up appointment will include the Patient Global Impression of Improvement (PGII), and a postoperative questionnaire eliciting overall satisfaction and development of new pelvic symptoms.

INTERVENTIONS:
Behavioral: Guided IMagery (GIM) — It's a program of directed thoughts and suggestions that guide your imagination to a relaxed and focused state.
  Arms: Guided IMagery (GIM)

SUMMARY:
We hypothesize that women who use GIM pre-operatively will feel more prepared for surgery, have less anxiety on the day of surgery and have higher satisfaction scores 6 weeks after surgery compared to women who undergo our routine pre-operative care.

DETAILED DESCRIPTION:
Guided imagery (GIM) is a program of directed thoughts and suggestions that guide your imagination to a relaxed and focused state. In clinical settings, it was originally found effective in treating patients suffering primarily from emotional or psychological issues by using descriptive language and the five senses to help the patient visualize their desired change or outcome (1, 2). More recently, GIM has been incorporated into chemotherapy and surgical settings. While it has not been conclusively found to improve outcomes, patients who received GIM reported feeling less anxious, less nausea following chemotherapy, slightly shorter surgical recovery times and a higher quality of life (3-8). While these studies suggest exciting prospects for the incorporation of GIM into the normal pre-op routine, we believe that they have left out one integral piece of the puzzle. We have previously found that patients who feel "unprepared" for surgery have less post-operative satisfaction (9). We propose that the stress and anxiety of the unknown during a patient's surgical experience can make them feel unprepared for surgery. Therefore, the same techniques that have been previously shown to decrease these symptoms in chemotherapy treatment and surgery should help patients feel more prepared, and therefore more satisfied with their surgical experience. This key finding would give sufficient support for the incorporation of GIM into the pre-op routine of any surgical patient, and may prove to be a successful vehicle for increasing the overall satisfaction of any hospital's patient population.

ELIGIBILITY:
Inclusion Criteria:

* routine vaginal or laparoscopic surgery for pelvic organ prolapse planned ≥ 1 week from enrollment
* a planned overnight hospital stay
* commitment to listen to a 15 minute audio Compact Disc daily
* proficiency in English.

Exclusion Criteria:

* Not having routine vaginal or laparoscopic surgery for pelvic organ prolapse planned ≥ 1 week from enrollment
* Not a planned overnight hospital stay
* Unable to commitment to listen to a 15 minute audio Compact Disc daily
* Not proficiency in English.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-06; Primary Completion 2016-02 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in patient satisfaction with urogynecological surgery when using GIM (questionnaire) | 6 weeks
  Women will report their satisfaction with their surgical experience 6 weeks after surgery using a 10-point Likert scale.

SECONDARY OUTCOMES:
Change in patient sense of preparedness when using GIM (questionnaire) | 6 weeks
  Preparedness will be measured at baseline, day of surgery, and 6 weeks after surgery to determine how GIM affected patient preparedness. It will be measured using a 10-point Likert scale
Change in patient anxiety about surgery when using GIM (questionnaire) | 6 week
  Patient anxiety will be measured at baseline, day of surgery and at 6 weeks post op to determine how GIM affected anxiety. It will be measured using the State-Trait Anxiety Inventory (STAI), which has been used extensively in research and clinical practice since its introduction in 1966 and is the most widely cited measure of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Mueller, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McKinney CH, Antoni MH, Kumar M, Tims FC, McCabe PM. Effects of guided imagery and music (GIM) therapy on mood and cortisol in healthy adults. Health Psychol. 1997 Jul;16(4):390-400. doi: 10.1037//0278-6133.16.4.390. PMID 9237092
- [Background] 1. Utay, J.; Miller, M. "Guided imagery as an effective therapeutic technique: a brief review of its history and efficacy research." Journal of Instructional Psychology, March 2006.
- [Background] Burns DS. The effect of the bonny method of guided imagery and music on the mood and life quality of cancer patients. J Music Ther. 2001 Spring;38(1):51-65. doi: 10.1093/jmt/38.1.51. PMID 11407965
- [Background] Walker LG, Walker MB, Ogston K, Heys SD, Ah-See AK, Miller ID, Hutcheon AW, Sarkar TK, Eremin O. Psychological, clinical and pathological effects of relaxation training and guided imagery during primary chemotherapy. Br J Cancer. 1999 Apr;80(1-2):262-8. doi: 10.1038/sj.bjc.6690349. PMID 10390006
- [Background] Holden-Lund C. Effects of relaxation with guided imagery on surgical stress and wound healing. Res Nurs Health. 1988 Aug;11(4):235-44. doi: 10.1002/nur.4770110405. PMID 3043570
- [Background] Fournier D, Boccara AC, Badoz J. Photothermal deflection Fourier transform spectroscopy: a tool for high-sensitivity absorption and dichroism measurements. Appl Opt. 1982 Jan 1;21(1):74-6. doi: 10.1364/AO.21.000074. PMID 20372403
- [Background] Halpin LS, Speir AM, CapoBianco P, Barnett SD. Guided imagery in cardiac surgery. Outcomes Manag. 2002 Jul-Sep;6(3):132-7. PMID 12134377
- [Background] Elkadry EA, Kenton KS, FitzGerald MP, Shott S, Brubaker L. Patient-selected goals: a new perspective on surgical outcome. Am J Obstet Gynecol. 2003 Dec;189(6):1551-7; discussion 1557-8. doi: 10.1016/s0002-9378(03)00932-3. PMID 14710061
- [Background] Barber MD, Walters MD, Bump RC. Short forms of two condition-specific quality-of-life questionnaires for women with pelvic floor disorders (PFDI-20 and PFIQ-7). Am J Obstet Gynecol. 2005 Jul;193(1):103-13. doi: 10.1016/j.ajog.2004.12.025. PMID 16021067
- [Background] Bump RC, Mattiasson A, Bo K, Brubaker LP, DeLancey JO, Klarskov P, Shull BL, Smith AR. The standardization of terminology of female pelvic organ prolapse and pelvic floor dysfunction. Am J Obstet Gynecol. 1996 Jul;175(1):10-7. doi: 10.1016/s0002-9378(96)70243-0. PMID 8694033
- [Background] 12. Spielberger, C.D., et al. State-Trait Anxiety Inventory (preliminary Test manual, Form B) Tallahassee, Florida: Florida State University, 1967
- [Background] Smith RC, Lay CD. State and trait anxiety: an annotated bibliography. Psychol Rep. 1974 Apr;34(2):519-94. No abstract available. PMID 4595041
- [Background] Pham T, Kenton K, Mueller E, Brubaker L. New pelvic symptoms are common after reconstructive pelvic surgery. Am J Obstet Gynecol. 2009 Jan;200(1):88.e1-5. doi: 10.1016/j.ajog.2008.08.010. Epub 2008 Oct 9. PMID 18845285